CLINICAL TRIAL: NCT05418452
Title: Efficacy of 1% Metformin Gel Mixed With PRF in Augmenting Narrow Ridge With Split-crest Technique and Implant Installation
Brief Title: Efficacy of 1% Metformin Gel Mixed With PRF in Augmenting Narrow Ridge
Acronym: MF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdelaziz Kamal Aboamo, assistant professor at AlAzharU department of Periodontology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 780/439
Record Dates: First submitted 2022-03-28; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Horizontal Ridge Deficiency
Keywords: implant; ridge split; metformin; PRF
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin (Experimental): will receive split-crest technique by ultrasonic bone surgery with implant placement and PRF mixed with 1% metformin gel
  Interventions: Drug: Metformin
- control (No Intervention): will receive split-crest technique by ultrasonic bone surgery with implant placement without gap filling.

INTERVENTIONS:
Drug: Metformin — metformin (MF), an antidiabetic agent, has been successfully used as a local drug delivery agent in periodontitis patients. Literature has suggested that MF possesses the osteogenic potential and induces the growth of osteoblast precursor cells. Therefore, several human studies have reported the use of MF alone or combined with PRF in the treatment of bony defects
  Arms: metformin

SUMMARY:
This study aimed to evaluate the efficacy of 1% metformin gel mixed with PRF, in horizontal ridge augmentation with the split-crest technique, for implant placement.

DETAILED DESCRIPTION:
Dental rehabilitation of edentulous patients with implants has become a common practice in the last few decades. Unfortunately, local conditions of some alveolar ridges of such patients may be challenging for implant placement. One of these conditions is a relevant horizontal deficit that may render dental implants difficult or impossible.

Several solutions are presented to overcome this challenge such as different guided bone regeneration (GBR) techniques and horizontal ridge split. However, these techniques have many shortages that may be overcome by the split crest technique (SCT).

SCT is a procedure for horizontal bone augmentation. It consists of splitting the vestibular and buccal cortical bone, displacing the vestibular cortical bone both in the maxilla or mandible, and separating from the bone marrow, creating a middle gap that is usually occupied mostly by the inserted implants. In such a procedure, ultrasonic bone surgery represents an advantageous alternative technique over conventional surgery using disks and chisels. The ultrasonic device can safely cut mineralized hard tissues such as bone with minor damage. Additionally, at the bone structural level, ultrasonic bone surgery may increase trabecular density as well as bone compression.

To enhance healing the remaining unoccupied space around the implant can be filled with biomaterials such as autologous bone grafts which are considered the gold stander, but unfortunately, site morbidity, as well as, utilizing more than one surgical site may limit its application. Alternatively, other bone substitutes including xenografts, alloplastic, and non-bone graft materials such as Platelet-Rich Fibrin (PRF) have been used in peri-implants space occupation.

PRF is a blood derivative in which platelets have a higher concentration above the baseline level. it can regulate inflammation and stimulate the immune process of chemotaxis. This natural material seems to accelerate the physiological wound healing with or without bone grafts to accelerate new bone formation. (6)In clinical practice, it has already been largely applied as an inexpensive carrier and way to obtain many growth factors (GFs) in physiological proportions. Hence, enhanced bone regeneration and favorable implant healing can be better achieved by using PRF as a graft around dental implants. Some authors reported that the use of PRF as a sole filling material during a simultaneous SCT and implantation stabilized a high volume of natural regenerated bone in the spaces unoccupied by the implants.

Lately, metformin (MF), an antidiabetic agent, has been successfully used as a local drug delivery agent in periodontitis patients. Literature has suggested that MF possesses the osteogenic potential and induces the growth of osteoblast precursor cells. Therefore, several human studies have reported the use of MF alone or combined with PRF in the treatment of bony defects Although PRF is an autogenous material obtained from a patient's blood and contains GFs which promote bone formation, its short time stability may not give it superiority over a commonly used bone graft like xenograft Adding a medical formula with osteogenic potential such as MF to PRF may add to its therapeutic performance and may present a graft material comparable to bone substitutes with the benefit of being cost-effective. Testing this hypothesis constitutes the primary aim of work in the present clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age 18-50) exhibiting initial insufficiently bone ridge.
2. Patients with good oral hygiene.
3. Free from systemic diseases that may influence the outcome of the therapy.

Exclusion Criteria:

1. Heavy smokers.
2. Patient treated by immunosuppressive chemotherapy or radiotherapy,
3. Allergy to any material or medication used in the study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Clinical parameter to measure difference | to detect change from baseline at time (immediately after implant insertion) and after 6 months.
  Implant stability (resonance frequency analysis)

SECONDARY OUTCOMES:
Radiological assessment to measure difference | to detect change from baseline (immediately after surgery), at time of loading (6 months), and 6 months after loading
  bone height

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar universty, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No